CLINICAL TRIAL: NCT07136077
Title: A Phase 2 Trial of Fruquintinib and Tislelizumab in ctDNA-defined Minimal Residual Disease in Colorectal Cancer After Completion of Adjuvant Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: BeiGene (Industry); Takeda Pharmaceutical Co. Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0696; NCI-2025-06047 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-08-18; First posted 2025-08-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Minimal Residual Disease; Adjuvant Chemotherapy; Colorectal Cancer; Fruquintinib; Tislelizumab; ctDNA
MeSH Terms: conditions — Neoplasm, Residual; Colorectal Neoplasms | interventions — tislelizumab; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase II: Treatment with Fruquintinib and Tislelizumab (Experimental): Treatment with Fruquintinib and Tislelizumab
  Interventions: Drug: Tislelizumab; Drug: Fruquintinib

INTERVENTIONS:
Drug: Tislelizumab — Given by IV
Drug: Fruquintinib — Give by PO

SUMMARY:
To find out if a combination of fruquintinib and tislelizumab can control CRC in patients who have received treatment for the disease but still have "positive" ctDNA tests for MRD (meaning there is evidence of MRD based on this test).

DETAILED DESCRIPTION:
Primary Objectives

• To determine the ctDNA clearance rate at 6 months in colorectal cancer participants with minimal residual disease following Fruquintinib and Tislelizumab therapy.

Secondary Objectives

* To determine the 3-month ctDNA clearance rates in colorectal cancer participants with minimal residual disease.
* To determine the disease-free survival (DFS) amongst colorectal cancer participants with minimal residual disease following Fruquintinib and Tislelizumab therapy.
* To determine the overall survival (OS) amongst colorectal cancer participants with minimal residual disease following Fruquintinib and Tislelizumab.
* To determine the safety and tolerability of Fruquintinib and Tislelizumab for the treatment of colorectal cancer participants with minimal residual disease.

ELIGIBILITY:
Eligibility Criteria

* Participants must have histologically or cytologically confirmed microsatellite stable (MSS) colorectal adenocarcinoma.
* Participants must have completed curative intent treatments of stages II, III, or IV colorectal cancer that must include ≥ 3 months of oxaliplatin containing chemotherapy.
* No evidence of radiographic disease within 28 days (before or after) a positive ctDNA assay.
* Participants must have minimal residual disease as defined by positive ctDNA assay (completed as standard-of-care at MD Anderson) such as Signatera. Participants may be identified for enrollment and followed with any Clinical Laboratory Improvement Amendments (CLIA)-certified ctDNA assay for MRD
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count of ≥1.0×109/L
  * Platelet count of ≥100×109/L
  * Hemoglobin ≥9 g/dL
  * Serum total bilirubin ≤1.5× upper limit of normal (ULN) (total bilirubin must be <3× ULN for participants with documented Gilbert's syndrome).
  * Participants without liver metastases must have ALT and AST ≤2.5× ULN; participants with liver metastases must have ALT and AST ≤5× ULN.
  * Urine protein ≤1+ by dipstick or 24-hour urine protein <1 g/24 hours. Participants with 2+ proteinuria by dipstick must undergo 24-hour urine collection to assess urine protein level.
  * Serum creatinine <1.5× ULN and creatinine creatinine clearance (CrCl) ≥30 mL/min per Cockcroft-Gault.
  * International normalized ratio (INR) and activated prothrombin time (aPTT) ≤1.5 ULN unless the participant is receiving anticoagulation therapy and INR and aPTT values are within the intended therapeutic range.
* ECOG performance status (PS) of 0 or 1.
* Age ≥ 18 years.
* Is able to understand and is willing to sign a written informed consent document.
* Is willing to utilize contraception. Women subjects of childbearing potential should agree to use highly effective contraception combined with an additional barrier method (eg, diaphragm, with a spermicide) while on study and for 4 months after last dose of study drug, and the same criteria are applicable to male subjects if they have a partner of childbirth potential. Male subject agrees to use a condom and not donate sperm while in this study and for 4 months after the last treatment.

Exclusion Criteria

* Has other concomitant active, invasive malignancies that may interfere with ctDNA analysis (known clonal hematopoesis of unknown potential allowed).
* Has serum electrolytes, potassium, calcium, or magnesium levels outside of the normal laboratory reference range which are clinically significant in the investigator's judgment.
* Has significant concomitant health conditions including but not limited to severe autoimmune or cardiovascular disorders that may interfere with participation in the study.
* Active autoimmune diseases or history of autoimmune diseases that may worsen or relapse per treating providers' evaluation.
* Has a persistent adverse event from previous treatment, except alopecia and neuropathy, greater than or equal to grade 2 of the Common Toxicity Criteria for Adverse Events (CTCAE) v. 5.0
* Systemic anti-neoplastic therapies or any investigational therapy within 4 weeks prior to the first dose of study drug, including chemotherapy, radical radiotherapy, hormonotherapy, biotherapy, and immunotherapy.
* Systemic small molecule-targeted therapies (eg, tyrosine kinase inhibitors) within 5 halflives or 4 weeks (whichever is shorter) prior to the first dose of study drug.
* Mean QT interval corrected by the method of Fridericia (QTcF) ≥480 ms.
* Has another disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition that investigators suspect may (a) prohibit use of the investigational product, (b) affect interpretation of study results, or (c) put the participant at undue risk of harm
* Has known hypersensitivity to the trial drugs or their excipients or is at risk of allergic of anaphylactic reaction to drug product according to the Investigator's judgement.
* Is pregnant or lactating.
* Is unable to take medication orally or has any other condition that investigators believe may affect absorption of the investigational product.
* Is receiving any other investigational agent.
* Any condition that requires systemic treatment with either corticosteroid (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days before the first dose of study drug(s), with the following exceptions:

  * Adrenal replacement (dose of ≤10 mg daily of prednisone or equivalent).
  * Topical, ocular, intra-articular, intranasal, or inhalational corticosteroid with minimal systemic absorption.
  * Short course (≤7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a non-autoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen)
* Live vaccine ≤28 days before the first dose of study drug(s). Seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.
* Known untreated or inadequately treated active hepatitis C, or chronic hepatitis B.
* Known untreated or inadequately treated human immunodeficiency virus (HIV) infection.
* Major surgery within 30 days before the first drug administration. Participants must have recovered adequately from the toxicity and/or complications from the intervention prior to the first dose of study drug(s).
* Prior allogeneic stem cell transplantation or organ transplantation.
* Any of the following cardiovascular risk factors:

  * Acute myocardial infarction ≤6 months before the first dose of study drug(s).
  * Heart failure meeting New York Heart Association Function Classification III or IV ≤6 months before the first dose of study drug(s)
  * Ventricular arrhythmia Grade ≥2 in severity ≤6 months before the first dose of study drug(s).
  * Cerebrovascular accident ≤12 months before the first dose of study drug(s).
  * Uncontrolled hypertension that cannot be managed by standard antihypertension medications, which is specified as systolic pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg. The participant must have blood pressures below both limits. Repeated assessments are permitted.
  * Syncope or seizure ≤28 days before the first dose of study drug(s).
* Received strong inducers of cytochrome P450, family 3, subfamily A (CYP3A) taken within 2 weeks (or 5 times the t1/2 of the drug, whichever is longer) prior to the first study treatment.
* Active gastrointestinal and duodenal ulcers, ulcerative colitis, and other gastrointestinal disease: other conditions that the investigator determines to possibly cause gastrointestinal bleeding, perforation, and other conditions; or prior gastrointestinal perforation or gastrointestinal fistula that has not recovered after surgical treatment.
* History or presence of clinically significant hemorrhage from any site (such as clinically significant melena, hematemesis, hemoptysis, fresh in stool) within 2 months before the screening.
* History of arterial thrombus within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Dasari, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org